CLINICAL TRIAL: NCT03353727
Title: Orthoptic Rehabilitation for Low Vision People With Innovative Mechanisms (Eye Tracker and Tactile Device)
Acronym: VISIONUM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of Financial support
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JGS_2016_25
Record Dates: First submitted 2017-10-25; First posted 2017-11-27 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2017-10

CONDITIONS: Low Vision
Keywords: Orthoptic rehabilitation; low vision; eye tracker; tactile device
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orthoptic rehabilitation (Experimental)
  Interventions: Other: Orthoptic rehabilitation

INTERVENTIONS:
Other: Orthoptic rehabilitation — Orthoptic rehabilitation using innovative mechanisms (eye tracker and tactile device) for low vision people

SUMMARY:
This project is working on orthoptic rehabilitation for low vision people. The aim of the project is to assess the interest and integration of this rehabilitation device used at home, in low-vision private practice and at the hospital. It leads to develop and evaluate an innovative device to integrate and adjust monitoring of patients according to their need and their progress, to create new interactions with the patient, enabling the orthoptist to stay in touch with his patient at home between rehabilitation sessions and to obtain a more fine and objective analysis of the exercises done by the patient.

Using an eye tracker and a digital tactile screen with data uploads allows the practitioner to observe the progress objectively. It also leads the patient to a better understanding of his/her visual behavior and of the effects of rehabilitation. Therefore, it will be easier to adopt better strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from visual impairment, with a need for visual rehabilitation
* Visual acuity (≤1.3 logMAR)
* Good knowledge of French language
* Informed consent of research

Exclusion Criteria:

* Medical treatment that may interfere with the study
* Degenerative diseases or any other diseases that may interfere with the study.
* Mini-Mental State Examination Score without visual item ≤ 20/25
* Pregnancy and lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
score assessing the feasibility of the rehabilitation | 18 months after inclusion
  System Usability Scale score

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Girmens, MD, Principal Investigator — Centre Hospitalier National d'Ophtalmologie des Quinze Vingts, Paris
Locations (3):
- France (3):
  - Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris
  - Fondation Hospitalière Sainte Marie, Paris
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris